CLINICAL TRIAL: NCT04861298
Title: Study to Investigate the Benefits of Dietary Supplement Quercetin for Early Symptoms of COVID-19
Brief Title: Study to Investigate the Clinical Benefits of Dietary Supplement Quercetin for Managing Early Mild Symptoms of COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 192/RC/KEMU
Record Dates: First submitted 2021-04-25; First posted 2021-04-27 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (SOC) (Active Comparator): This arm will receive the standard of care (SOC) for COVID-19 as per the hospital guidelines.
  Interventions: Drug: standard of care for COVID-19 as per the hospital guidelines
- Quercetin (Experimental): This arm will receive standard of care + oral Quercetin for two weeks
  Interventions: Drug: standard of care for COVID-19 as per the hospital guidelines; Dietary Supplement: Quercetin Phytosome (QP)

INTERVENTIONS:
Drug: standard of care for COVID-19 as per the hospital guidelines — Hospital standard of care treatment for COVID-19
Dietary Supplement: Quercetin Phytosome (QP) — Daily dose of 600 mg of Quercetin for 1st week and then 400 mg for the 2nd week
  Arms: Quercetin

SUMMARY:
Quercetin is a flavonoid dietary supplement that occurs in many edible fruits and vegetables. It has remarkable antioxidant, anti-inflammatory, immunoprotective and antiviral properties. It is widely used to boost the body immune system against infections and keeping healthy life-style. The purpose of the present study is to investigate the potential benefits of quercetin for preventing COVID-19 disease progression and symptoms improvement in the early stage of infection.

DETAILED DESCRIPTION:
The strong antioxidant and anti-inflammatory properties of quercetin are closely related to its effective fight against a variety of disease conditions related to inflammation, including: viral infections, allergies, asthma, hay fever, arthritis, respiratory diseases, "hardening of the arteries" (atherosclerosis), high cholesterol, heart disease and circulation problems, insulin resistance and diabetes, eye-related disorders, including cataracts, stomach ulcers, cognitive impairment, gout, cancer, chronic fatigue syndrome, inflammation of the prostate, bladder, and ovaries, chronic infections of the prostate, skin disorders, including dermatitis and hives. Quercetin can help stop damaging particles in the body known as free radicals, which damages the cells by natural oxidation processes. It can also reduce the expression of inflammatory genes in the cells.

Quercetin has been shown to be effective against broad range of viruses including human respiratory syncytial virus (hRSV), rhinovirus, echovirus, coxsackievirus, poliovirus, parainfluenza type 3, Herpes Simplex Virus-1, cytomegalovirus, SARS-CoV-1, dengue virus, and Hepatitis C virus.

The purpose of the present study is to investigate the potential benefits of quercetin for preventing COVID-19 disease progression and improving symptoms in the early stage of infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18 years of age or older, of either gender
* Patients must be tested positive for SARS-CoV-2 by RT-PCR
* Patients must exhibit typical symptoms of COVID-19 disease at screening such as fever, fatigue, a dry and contagious cough, loss of appetite, body aches, shortness of breath, mucus or phlegm, sore throat, headache, chills, sometimes with shaking, loss of smell or taste, congestion or runny nose, nausea, or vomiting, diarrhea, muscular pain etc.
* Patients must be in the early stage of COVID-19 disease who do not require hospitalisation at the time of screening
* Patients must be under the care of a Physician for diagnosis of COVID-19
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with proven hypersensitivity or allergic reaction to quercetin
* Patients with known chronic kidney disease with estimated creatinine clearance < 50 mL/minute or need for dialysis
* Patients who are severely hypotensive defined as needing hemodynamic pressors to maintain blood pressure
* Patients with moderate or severe thrombocytopenia (platelet count <100 × 10⁹/L);
* Pregnant patients
* Patients declining to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-08-29 (Actual); Study Completion 2021-08-29 (Actual)

PRIMARY OUTCOMES:
Testing negative for SARS-CoV-2 by RT-PCR with symptoms improvement | From day 1 to day 14

SECONDARY OUTCOMES:
Percentage of subjects that require hospitalisation | From day 1 to day 14
Improvement in CRP | From day 1 to day 14
Improvement in D-Dimers | From day 1 to day 14
Improvement in LDH | From day 1 to day 14
Improvement in Ferritin | From day 1 to day 14
Improvement in CBC | From day 1 to day 14

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Di Pierro F, Khan A, Iqtadar S, Mumtaz SU, Chaudhry MNA, Bertuccioli A, Derosa G, Maffioli P, Togni S, Riva A, Allegrini P, Recchia M, Zerbinati N. Quercetin as a possible complementary agent for early-stage COVID-19: Concluding results of a randomized clinical trial. Front Pharmacol. 2023 Jan 13;13:1096853. doi: 10.3389/fphar.2022.1096853. eCollection 2022. PMID 36712674